CLINICAL TRIAL: NCT02334943
Title: Immune Activation in HIV-1 Infected Patients Under AntiRetroviral Treatment: Etiologic Factors, Forms and Potential Association With Chronic Comorbidities Unrelated to Immune Deficiency.
Brief Title: Immune Activation in HIV-1 Infected Patients Under AntiRetroviral Treatment
Acronym: ACTIVIH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 9187
Record Dates: First submitted 2014-07-22; First posted 2015-01-08 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Immune Deficiency; HIV-related Gut Disease - Cause Unknown; Activation of Latent Virus; Other Diagnoses, Comorbidities, and Complications
Keywords: Immune Activation; HIV-1 infected subjects; Undetectable viral load; Causes of Immune Activation in HIV-1 infected patients; Forms of Immune Activation; Emergent non-AIDS related comorbidities
MeSH Terms: conditions — Immunologic Deficiency Syndromes | interventions — Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Treated HIV-1 infected patients (Experimental): Treated HIV-1 infected patients for Blood test
  Interventions: Biological: Blood test
- No treated HIV-1 infected patients (Experimental): No treated HIV-1 infected patients for Blood test
  Interventions: Biological: Blood test
- Healthy witness (Experimental): Healthy witness for Blood test
  Interventions: Biological: Blood test

INTERVENTIONS:
Biological: Blood test — Blood test

SUMMARY:
Immune Activation persists in HIV-1 infected patients despite efficient antiretroviral treatment. This immune activation is responsible for immune deficiency as well as for non-AIDS related comorbidities, such as non-alcoholic Fatty liver disease, metabolic syndrome or osteoporosis. The goal of this observational transversal multicentric study is to establish the etiologic factors of persistent immune activation in treated HIV-1 infected patients (persistent de novo infection of T CD4+ cells, microbial translocation, active coinfections, immunosenescence, T CD4+ cells lymphopenia, Treg deficiency), its different forms ( activation of T CD4+ cells, T CD8+ cells, B cells, NK cells, monocytes, granulocytes, platelets, endothelial cells or general inflammation) and the potential correlation between causes, forms of immune activation and emergent comorbidities (kidney, bone or liver dysfunction, metabolic syndrome).

DETAILED DESCRIPTION:
Immune Activation persists in HIV-1 infected patients despite efficient antiretroviral treatment. This immune activation is responsible for immune deficiency as well as for non-AIDS related comorbidities, such as non-alcoholic Fatty liver disease, metabolic syndrome or osteoporosis. The goal of this observational transversal multicentric study is to establish the etiologic factors of persistent immune activation in treated HIV-1 infected patients (persistent de novo infection of T CD4+ cells, microbial translocation, active coinfections, immunosenescence, T CD4+ cells lymphopenia, Treg deficiency), its different forms ( activation of T CD4+ cells, T CD8+ cells, B cells, NK cells, monocytes, granulocytes, platelets, endothelial cells or general inflammation) and the potential correlation between causes, forms of immune activation and emergent comorbidities (kidney, bone or liver dysfunction, metabolic syndrome). These correlations could highlight physiopathologic mechanisms relating a specific cause of immune activation, activation of a specific subpopulation of immune cells and a comorbidity. Physiopathologic mechanisms could then be tested in vitro and lead into new therapeutic tracks of immune activation secondary to HIV-1 or to the natural ageing process.

ELIGIBILITY:
Inclusion criteria:

* Age > or = 45 years
* HIV-1 infection
* Number of T CD4+ lymphocytes before antiretroviral treatment < 350 cells/mm3
* Current number of T CD4+ lymphocytes > 200 cells / mm3 for 6 moths before inclusion
* Efficient and well tolerated antiretroviral treatment for more than 24 months
* HIV-1 viral load < 50 copies/ml for more than 24 months before inclusion
* Patient able to understand the nature, the objective and the methods of the study
* Patient having signed the informed consent
* Affiliation to French Social Security System

Exclusion criteria:

* Patient having a current evidence of II to IV rank of the ANRS scale clinical condition
* Patient having a current evidence of III to IV rank of the ANRS scale biological condition
* Patient has a current evidence of an active coinfection
* Patient has a current (active) diagnosis of acute hepatitis due to any cause. Patients with chronic hepatitis, including chronic hepatitis B and/or C, may enter the study as long as they have stable liver function tests and undetectable viral load of hepatitis B and/or C
* Patient has a cirrhosis
* Patient presents with a non infectious pathology that might give immune modifications
* Patient using immuno-modulator therapy or chemotherapy
* Patient is currently participating or has participated in a study (within the exclusion period defined by this study)
* Patient is pregnant or breastfeeding

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2015-03; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Infection of novo persistent | Infection of novo persistent the day of inclusion
  Etiologic factors of persistent immune activation in treated HIV-1 infected patients (obstinacy of the infection of new cells T CD4 +, microbial translocation, active coinfection, immunosenescence, lymphopenia T CD4 +, deficit in lymphocytes Treg) on a day: the day of the inclusion

SECONDARY OUTCOMES:
Microbial translocation | Microbial translocation the day of inclusion
  Microbial translocation (DNA bacterial plasma derivative)
Diagnosis immunizing activation | Diagnosis immunizing activation the day of inclusion
  Activation T CD4 and T CD8, B, NK

OTHER OUTCOMES:
No immunological response to treatment | No immunological response to treatment the day of inclusion
  Measurement of circulating CD4 +
Renal Review | Renal Review the day of inclusion
  Estimated glomerular filtration rate, Na / K / Cl / alkaline reserve, blood uric acid, typing with proteinuria, albuminuria, creatinine, phosphorus reabsorption, urine dipstick
Bone balance | Bone balance the day of inclusion
  Determination of Calcium and phosphate levels in fasting, PTH, TSH, 25hydroxy vitamin D, testosterone (male), estradiol (female)
Metabolic syndrome assessment | Metabolic syndrome assessment the day of inclusion
  Metasting blood glucose, HbA1c, triglycerides, LDL cholesterol, HDL cholesterol

CONTACTS AND LOCATIONS:
Overall Officials: JACQUES REYNES, PU PH, Principal Investigator — Univerty Hospital Montpellier
Locations (1):
- University hospital Montpellier, Montpellier, France